CLINICAL TRIAL: NCT06897020
Title: Evaluation of Child and Parental Satisfaction of Bioflx Crowns Compared to Zirconia Crowns on Primary Molars
Brief Title: Child and Parental Satisfaction of Bioflx Crowns Compared to Zirconia Crowns in Primary Molars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Razan Adil Yousif Ahmed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPS - Bioflx Vs ZR
Record Dates: First submitted 2025-03-20; First posted 2025-03-26 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Carious Primary Molars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- (Group A: Performed Bioflx crowns) (Experimental): Bioflx Crowns, claimed to be the first flexible, durable, and aesthetic preformed crowns for primary molars. Bioflx are monochromatic, metal-free, tooth-colored crowns made from a high-strength resin polymer used in the medical device industry, offering strength, flexibility, and durability.These crowns are autoclavable and are claimed to require similar tooth preparation as SSCs.
  Interventions: Other: (Group A: Bioflx crowns)
- (Group B: Preformed zirconia crown) (Experimental): Zirconia crowns brought a concept shift in esthetics of crowns; they are the most esthetic option available for treating primary molars. These crowns are resilient, tooth-colored, and highly polished. Zirconia crowns provide a more natural, tooth-colored alternative, making them a preferred option in cases where aesthetics is a priority.
  Interventions: Other: (Group B: Preformed Zirconia crown

INTERVENTIONS:
Other: (Group A: Bioflx crowns) — prepartion:1.The mesiodistal width of the tooth will be measured using calipers and a closely fitted crown will be selected based on the measurements.
  2.The tooth will be prepared similarly to stainless steel crowns (SSCs): • Occlusal reduction of approximately 1-1.5 mm will be done using a diamond bur.Mesial and distal reduction of no more than 1 mm will be performed using a No. 169L diamond bur.Depending on the tooth anatomy, either no buccal and lingual reduction will be needed, or a minimal reduction will be done. 3.All sharp line angles and corners will be smoothed to ensure proper crown fit. 4.The crown will be checked for proper fit before cementation. It will be positioned to extend 1 mm below the gingival margin. 5.The crown will be cemented using luting glass ionomer cement (GIC). The crown will be held with firm, constant pressure until the cement sets initially.
  6.The marginal fit will be evaluated, and necessary adjustments will be made. 7.The occlusion will be checked.
  Arms: (Group A: Performed Bioflx crowns)
Other: (Group B: Preformed Zirconia crown — 1. Crown Selection: The mesiodistal dimension of the corresponding tooth will be measured . to select the appropriate size.
  2. Occlusal Reduction: The marginal ridge of adjacent teeth will be used as a reference point and a 1.5-2 mm of occlusal reduction will be performed to allow proper crown seating.
  3. Bucco-Lingual Reduction: The bucco-lingual wall will be reduced by approximately 1-1.5 mm using a flame-shaped diamond bur.
  4. Interproximal Reduction: 1mm of interproximal reduction will be performed using a flame-shaped diamond bur such as a .368 or .330tapered carbide bur.
  5. Feather Margin Preparation: Subgingival reduction of 1-2 mm will be done using a flame-shaped diamond bur, creating a feathered margin to achieve a passive fit.
  6. Trial Fitting of the Crown: The crown will be tried in to ensure proper adaptation. until the crown fits passively and extends sub gingivally by 1-2 mm wit.
  7. Glass ionomer cement will be used for cementation.
  Arms: (Group B: Preformed zirconia crown)

SUMMARY:
The goal of this clinical trial is to evaluate the child and parents satisfaction of Bioflx crowns compared to zirconia crowns in the restoration of primary molars. The main question[s] it aims to answer : Is there a difference in the child and parents satisfaction levels between BioFlx crowns and zirconia crowns in the restoration of primary molars?" The study will also assess the clinical performance of both types of crowns in terms of Retention, occlusal wear, gingival health, as well as preparation time.

DETAILED DESCRIPTION:
The management of severely decayed primary teeth in pediatric dentistry often requires the use of crowns to restore function and aesthetics. Traditional stainless-steel crowns (SSCs) have been widely used due to their durability and cost-effectiveness; however, their metallic appearance and lack of aesthetic appeal have prompted the development of alternative materials such as zirconia and Bioflx crown. Zirconia crowns are recognized for their superior aesthetics and biocompatibility, making them a preferred choice for parents who prioritize appearance. However, they can present challenges in terms of retention, preparation requirements, and cost. Bioflx crowns, a newer material in pediatric dentistry, aim to combine aesthetic appeal with flexibility and improved adaptability to tooth anatomy. Despite their growing popularity, limited research directly compares the child and parental satisfaction between zirconia and Bioflx crowns. It remains unclear which material offers the best balance of functional, aesthetic, and patient-centered outcomes.This gap in knowledge hinders evidence-based decision-making when selecting crowns for pediatric patients. Zirconia crowns have gained prominence in pediatric dentistry as an alternative to stainless steel crowns for primary molars. While SSCs have long been valued for their durability and ease of placement, their metallic appearance often presents an aesthetic concern for parents and patients. Zirconia crowns provide a more natural, tooth-colored alternative, making them a preferred option in cases where aesthetics is a priority. One of the main advantages of zirconia crowns is their biocompatibility, as they demonstrate lower plaque accumulation and gingival inflammation. Additionally, zirconia crowns offer superior mechanical properties, including high flexural strength and excellent fracture resistance, making them a long-lasting restorative option. Their wear resistance further supports their use in pediatric patients, particularly those with heavy occlusal forces. This study stems from the need to bridge the gap in current research regarding the satisfaction and the effectiveness associated with Bioflx crowns. Understanding whether Bioflx crowns offer superior aesthetic and functional outcomes compared to Zirconia crowns could influence clinical decision-making in pediatric dentistry. This is especially relevant as parents increasingly seek restorations that provide both durability and a natural appearance for their children.

ELIGIBILITY:
Inclusion Criteria:

* The Inclusion criteria:

  1. Children aged four to eight years old who are appearing healthy and free of any systemic disease according to parental history.
  2. Frankl's positive and definitely positive children.
  3. Children whose parent or guardian are willing to sign an informed consent.
  4. Children whose parent or guardian are willing to comply with follow-up visits.
  5. Primary molars indicated for crowns. • Exclusion criteria:

  <!-- -->

  1. Children with

Exclusion Criteria:

* The Exclusion criteria:

  1. Children with poor oral hygiene that may contribute to higher plaque levels and affect the clinical outcomes of the crown restorations.
  2. Children with history of allergies; Known allergies to dental local anesthesia or to the materials used in Bioflx crowns.
  3. Child with parafunctional habits.
  4. Molars with severe structural loss that may compromise crown retention.
  5. Presence of malocclusion such as crossbite or scissor bite.
  6. Primary molar with root caries.
  7. Primary molar with root resorption or furcation involvement.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-26 (Estimated)

PRIMARY OUTCOMES:
Child and Parents Satisfaction | [Time Frame: T (Time): 6months interval T0: 0T1: 3month T2: 6month]
  Method of Measurement:
  * 5-Point likert's scale unites of measurement:
    1. Very Happy.
    2. Happy.
    3. Neither.
    4. Unhappy.
    5. Very Unhappy.
  * Questionnaire:Ordinary or N/A existing validated tool.

SECONDARY OUTCOMES:
Retention | [Time Frame: follow-up:T (Time): 6months interval T0: 0 T1: 3month T2: 6month]
  Measure by Modified United States Public Health System criteria:
  Alpha: Intact. Bravo:Chipped/loss of material. Charlie: Complete loss of crown.
Occlusal wear of crown | [Time Frame: T (Time): 6months interval T0: 0 T1: 3 month T2: 6month]
  Measure by Modified United States Public Health System criteria:
  Alpha: Occlusal surface intact. Bravo: Wear of occlusal surface without tooth surface exposure. Charlie: Wear of occlusal surface with exposure.
Gingival health | [Time Frame: T (Time): 6months interval T0: 0 T1: 3month T2: 6month]
  Measure by: Gingival index:
  0: healthy gum.
  1. mild discoloration and edematous gingiva no bleeding on probing.
  2. red oedematous and shiny gingiva bleeding on probing.
  3. red oedematous and ulceration gingiva spontaneous bleeding.
Preparation time | [Time Frame: baseline]
  Measure by :Stopwatch per minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Prof.Dr. Manal Ahmed Elshiekh, Ph.D, Study Director — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo University., Giza, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mathew MG, Roopa KB, Soni AJ, Khan MM, Kauser A. Evaluation of Clinical Success, Parental and Child Satisfaction of Stainless Steel Crowns and Zirconia Crowns in Primary Molars. J Family Med Prim Care. 2020 Mar 26;9(3):1418-1423. doi: 10.4103/jfmpc.jfmpc_1006_19. eCollection 2020 Mar. PMID 32509626
- [Background] Patil AS, Jain M, Choubey S, Patil M, Chunawala Y. Comparative evaluation of clinical success of Stainless Steel and Bioflx crowns in primary molar - A 12 month split mouth prospective randomized clinical trial. J Indian Soc Pedod Prev Dent. 2024 Jan 1;42(1):37-45. doi: 10.4103/JISPPD.JISPPD_484_23. Epub 2024 Apr 15. PMID 38616425